CLINICAL TRIAL: NCT01966367
Title: CD34+ Stem Cell Selection for Patients Receiving a Matched or Partially Matched Family or Unrelated Adult Donor Allogeneic Stem Cell Transplantation for Non-Malignant Disease
Brief Title: CD34+ (Non-Malignant) Stem Cell Selection for Patients Receiving Allogeneic Stem Cell Transplantation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Diane George (Other)
Responsible Party: Sponsor-Investigator, Diane George, Assistant Professor of Pediatrics, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAL0156
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Bone Marrow Failure Syndrome; Severe Aplastic Anemia; Severe Congenital Neutropenia; Amegakaryocytic Thrombocytopenia; Diamond-Blackfan Anemia; Schwachman Diamond Syndrome; Primary Immunodeficiency Syndromes; Acquired Immunodeficiency Syndromes; Histiocytic Syndrome; Familial Hemophagocytic Lymphocytosis; Lymphohistiocytosis; Macrophage Activation Syndrome; Langerhans Cell Histiocytosis (LCH); Hemoglobinopathies; Sickle Cell Disease; Sickle Cell-beta-thalassemia
Keywords: Unrelated donor transplant; Haploidentical donor transplant; Peripheral blood stem cell transplantation; CD34+ selection; Non-malignant disease; Bone marrow failure syndrome; Severe Aplastic Anemia; Severe Congenital Neutropenia; Amegakaryocytic Thrombocytopenia; Diamond-Blackfan Anemia; Schwachman Diamond Syndrome; Primary Immunodeficiency Syndrome; Acquired Immunodeficiency Syndrome; Histiocytic Syndrome; Familial Hemophagocytic Lymphocytosis; Lymphohistiocytosis; Macrophage Activation Syndrome; Langerhans Cell Histiocytosis (LCH); Hemoglobinopathies; Sickle Cell Disease; Sickle Cell-beta-thalassemia
MeSH Terms: conditions — Bone Marrow Failure Disorders; Anemia, Aplastic; Neutropenia, Severe Congenital, Autosomal Recessive 3; Anemia, Diamond-Blackfan; Shwachman-Diamond Syndrome; Primary Immunodeficiency Diseases; Acquired Immunodeficiency Syndrome; Histiocytosis; Lymphohistiocytosis, Hemophagocytic; Macrophage Activation Syndrome; Histiocytosis, Langerhans-Cell; Hemoglobinopathies; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CliniMACS PLUS followed by chemotherapy (Experimental): Patients will receive a pre-transplant conditioning regimen of Busulfan Fludarabine and Alemtuzumab. For patients with pre-transplant hepatic dysfunction, Melphalan will be substituted for the Busulfan. For patients receiving a second transplant or a "boost", pre-transplant conditioning based on the clinical condition of the patient will be determined by the Principal Investigator and the patient's bone marrow transplantation (BMT) physician. The donor peripheral blood stem cells will undergo CD34+ selection (Biological/Vaccine: CD34 Stem Cell Selection Therapy). The CliniMACS (PLUS) Reagent System will be used to remove T-cells from the peripheral blood stem cell transplant in order to decrease the risk of acute and chronic graft versus host disease (GVHD).
  Interventions: Biological: CD34 Stem Cell Selection Therapy

INTERVENTIONS:
Biological: CD34 Stem Cell Selection Therapy — The CliniMACS (PLUS) Reagent System (Miltenyi CliniMACS CD34+ Cell Selection Device) will be used to remove T-cells from the peripheral blood stem cell transplant in order to decrease the risk of acute and chronic graft versus host disease (GVHD).

SUMMARY:
This study's goal is to determine the frequency and severity of acute graft versus host disease, to evaluate incidence of primary and secondary graft rejection, to assess event free survival and overall survival, to determine the time to neutrophil and platelet engraftment, to determine the time to immune reconstitution (including normalization of T, B and natural killer (NK) cell repertoire and Immunoglobulin G production), and to establish the incidence of infectious complications including bacterial, viral, fungal and atypical mycobacterial and other infections following CD34+ selection in children, adolescents and young adults receiving an allogeneic peripheral blood stem cell transplant from a family member or unrelated adult donor for a non-malignant disease.

DETAILED DESCRIPTION:
Graft-versus-host disease (GVHD) is a condition that results from a reaction of transplanted donor T-lymphocytes against the body and organs of the patient receiving the transplanted cells. There are two forms: acute (early) and chronic (late). Acute GVHD may produce skin rashes, liver disease, diarrhea, and an increased risk of infection. Chronic GVHD can appear in patients without prior acute GVHD. Chronic GVHD may also produce skin rashes, liver disease, diarrhea and an increased risk of infection. GVHD can make patients very sick, and have GVHD can make it more likely that patients will not survive their transplant. In this study, the investigators are offering to treat the donor peripheral blood stem cells in the hope that it will make it less likely for the patient who receives them from having GVHD.

Patients on this study are being offered an experimental treatment involving the use of the CliniMACS® Reagent System (Miltenyi Biotec, Germany), a CD34+ selection device to remove T-cells from the peripheral blood stem cell transplant in order to decrease the risk of acute and chronic GVHD. CD34+ stem cells are selected from the donor's peripheral blood stem cells. In doing this, T-cells are also removed. T-cells are the cells which are responsible for graft versus host disease (GVHD). This study is a clinical trial for patients diagnosed with a non-malignant disease who will receive a peripheral blood stem cell transplant. Patients with the following types of non-malignant diseases can participate in this study: Bone marrow failure syndromes (including Severe Aplastic Anemia, Severe Congenital Neutropenia, Amegakaryocytic Thrombocytopenia (Kostmann's Syndrome), Diamond-Blackfan Anemia, Schwachman Diamond Syndrome, Primary Immunodeficiency Syndromes, Acquired Immunodeficiency Syndromes, and Histiocytic Disorders) and Hemoglobinopathies (including Sickle Cell Anemia and Sickle/Beta Thalassemia). Patients on this study will be given standard transplant therapy with either high doses of chemotherapy drugs or lower doses of chemotherapy drugs, depending on their disease. Diseases within each disease group will receive chemotherapy that is standard for that condition.

Some patients on this study will receive an allogeneic stem cell transplant (AlloSCT) from a matched related donor. If a patient does not have a matched related donor, a bone marrow search will be done at all of the bone marrow banks in the world. The patient will then go on to receive an AlloSCT from either a partially matched family member or an unrelated adult stem cell transplant donor. The transplanted cells will allow all the normal parts of the patient's blood system to recover. The experimental portion of this treatment involves the use of a Miltenyi CliniMACS CD34+ selection device to remove T-cells from the peripheral blood stem cell transplant in order to decrease the risk of acute and chronic GVHD. CD34+ stem cell selection AlloSCT has been studied in adults with the malignant and non-malignant disease with successful engraftment and has shown some improvement in GVHD. It is unknown if CD34+ stem cell selection will work to prevent severe GVHD in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* General Eligibility (All Patients)

  * Patient must be < or = 40 years of age. Patients with sickle cell anemia must be at least 2 years of age.
  * Patient or the patient's legally authorized guardian must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign an informed consent in accordance with the institutional policies approved by the U.S. Department of Health and Human Services.
  * Approval for the use of this treatment protocol by the individual institution's Human Rights Committee must be obtained, in accordance with the institutional assurance policies of the U. S. Department of Health and Human Services.
  * Human leukocyte antigen (HLA) typing will be performed by high-resolution molecular DNA typing for HLA Class I A, B, and C and HLA Class II DRB1 and DQB1 alleles.

    * Unrelated donor: An 8/10, 9/10 or 10/10 matched unrelated adult donor (MUD) will be required for study entry.
    * Related Donor: A 5/10, 6/10, 7/10, 8/10, 9/10 or 10/10 matched (or partially matched) family donor will be required for study entry.
  * Non-malignant Disorders per protocol.
  * Hemoglobinopathies per protocol.
  * Requirement for CD34+ stem cell selection for a second infusion of stem cells following an allogeneic stem cell transplant from a related or unrelated adult donor.
* Additional eligibility for patients with non-malignant disorders receiving myeloablative conditioning

  * Adequate renal function as determined by the institutional normal range.
  * Adequate liver function per protocol.
  * Adequate cardiac function defined by radionucleotide angiogram or echocardiogram.
  * Adequate pulmonary function by pulmonary function test. For children who are uncooperative, no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry >94% on room air.
* Additional eligibility for patients with non-malignant disorders receiving reduced intensity conditioning

  * Adequate renal function as determined by the institutional normal range.
  * Adequate liver function per protocol.
  * Adequate cardiac function per protocol.
  * Adequate pulmonary function per protocol.

Exclusion Criteria:

* Patients with documented uncontrolled infection at the time of study entry are not eligible.
* Pregnancy/Breast-Feeding Females who are pregnant or breast feeding at the time of study entry are not eligible.

  -- The following additional exclusion criteria for patients with sickle cell anemia the following exclusion criteria also apply
* Patients with bridging fibrosis or cirrhosis of the liver.
* Uncontrolled bacterial, viral or fungal infection in the past month.
* Seropositivity for HIV.
* Patients who have received prior hematocrit (HCT) within three months of enrollment for reduced intensity regimen and within six months for myeloablative regimen/reduced toxicity regimens.

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute graft versus host disease (GVHD) | 100 days
  Determine the incidence and severity of acute GVHD.

SECONDARY OUTCOMES:
Incidence of primary graft failure | 1 year
  Quantify the incidence of primary and secondary graft failure.
Survival Rate | 5 years
  To assess event free survival and overall survival
Time to neutrophil and platelet engraftment | 1 year
  To determine the time to neutrophil and platelet engraftment
Time to immune reconstitution | 2 years
  To determine the time to immune reconstitution (including normalization of T, B and NK cell repertoire and Immunoglobulin G production)
Incidence of infectious complications | 2 years
  To establish the incidence of infectious complications including bacterial, viral, fungal and atypical mycobacterial and other infections
Incidence of secondary graft failure | 1 year
  Quantify the incidence of primary and secondary graft failure.

CONTACTS AND LOCATIONS:
Overall Officials: Diane George, MD, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital, New York-Presbyterian, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided